CLINICAL TRIAL: NCT05264337
Title: Lymphedema in the Lower Extremities After Urologic Surgery With Lymph Node Dissection
Brief Title: Lymphedema After Urologic Surgery
Status: Recruiting | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021-04840
Record Dates: First submitted 2022-02-03; First posted 2022-03-03 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Urinary Bladder Neoplasms; Prostatic Neoplasms; Testicular Neoplasms; Penile Cancer
Keywords: Lymphedema; Lymph Node Excision
MeSH Terms: conditions — Urinary Bladder Neoplasms; Prostatic Neoplasms; Testicular Neoplasms; Penile Neoplasms; Lymphedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Radical Cystectomy: Patients undergoing radical cystectomy with pelvic lymph node dissection for urinary bladder cancer
  Interventions: Other: Self-reported lymphedema; Other: Dielectric constant ratio; Other: Limb volume
- Radical Prostatectomy: Patients undergoing radical prostatectomy with pelvic lymph node dissection for prostate cancer
  Interventions: Other: Self-reported lymphedema
- Retroperitoneal: Patients undergoing retroperitoneal lymph node dissection for testicular cancer
  Interventions: Other: Self-reported lymphedema
- Other: Patients undergoing other urologic surgery with lymph node dissection of inguinal, iliacal or retroperitoneal lymph nodes
  Interventions: Other: Self-reported lymphedema

INTERVENTIONS:
Other: Self-reported lymphedema — Lymphedema as reported by LymQOL questionnaire.
Other: Dielectric constant ratio — Measurement of percentage tissue water content of lower extremities by dielectric constant ratio measured by MoistureMeter D.
  Groups: Radical Cystectomy
Other: Limb volume — Measurement of lymphedema by limb volume of lower extremities by multiple measurements of circumference.
  Groups: Radical Cystectomy

SUMMARY:
Lymphedema of the extremities is common after lymph node surgery in treating several forms of cancer, e.g., breast cancer. However, very little is known of the occurrence of lymphedema of the lower extremities after urologic surgery with lymph node dissection. This project aims to describe the frequency and grade of lymphedema arising after urologic surgery, using the Lymphedema Quality of Life Questionnaire (LymQOL), Delfin MoistureMeter D, and lower limb volume measurements.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing urologic surgery with lymph node dissection

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing urologic surgery that includes lymph node dissection
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-03-14 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with self-reported lymphedema at 12 months | 12 months after surgery
  Frequency and grade of self-reported swelling of the lower extremities as graded by LymQOL questionnaire
Number of patients with self-reported lymphedema at 24 months | 24 months after surgery
  Frequency and grade of self-reported swelling of the lower extremities as graded by LymQOL questionnaire
Change in tissue water content measured by MoistureMeterD Compact at 12 months | 12 months after surgery
  Percent tissue water content calculated from the dielectric constant as measured by MoistureMeterD Compact
Change in tissue water content measured by MoistureMeterD Compact at 24 months | 24 months after surgery
  Percent tissue water content calculated from the dielectric constant as measured by MoistureMeterD Compact
Change in lower limb volume calculated by measuring the circumference of the lower extremities at 12 months | 12 months after surgery
Change in lower limb volume calculated by measuring the circumference of the lower extremities at 24 months | 24 months after surgery

SECONDARY OUTCOMES:
Number of patients with self-reported lymphedema at 1 month | 1 month after surgery
  Frequency and grade of self-reported swelling of the lower extremities as graded by LymQOL questionnaire
Number of patients with self-reported lymphedema at 3 months | 3 months after surgery
  Frequency and grade of self-reported swelling of the lower extremities as graded by LymQOL questionnaire
Number of patients with self-reported lymphedema at 6 months | 6 months after surgery
  Frequency and grade of self-reported swelling of the lower extremities as graded by LymQOL questionnaire
Change in tissue water content measured by MoistureMeterD Compact at 1 month | 1 month after surgery
  Percent tissue water content calculated from the dielectric constant as measured by MoistureMeterD Compact
Change in tissue water content measured by MoistureMeterD Compact at 3 months | 3 months after surgery
  Percent tissue water content calculated from the dielectric constant as measured by MoistureMeterD Compact
Change in tissue water content measured by MoistureMeterD Compact at 6 months | 6 months after surgery
  Percent tissue water content calculated from the dielectric constant as measured by MoistureMeterD Compact
Change in lower limb volume calculated by measuring the circumference of the lower extremities at 1 month | 1 month after surgery
  Measurements of circumference every 6 cm along the lower limbs.
Change in lower limb volume calculated by measuring the circumference of the lower extremities at 3 month | 3 month after surgery
  Measurements of circumference every 6 cm along the lower limbs.
Change in lower limb volume calculated by measuring the circumference of the lower extremities at 6 month | 6 month after surgery
  Measurements of circumference every 6 cm along the lower limbs.

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Kjölhede, MD, PhD, Principal Investigator — Sahlgrenska University Hospital, Gothenburg University
Locations (2):
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Örebro University Hospital, Örebro

IPD SHARING:
Plan to Share IPD: No